CLINICAL TRIAL: NCT01174316
Title: Autotitrating Non-invasive Ventilation (NIV) Versus Standard NIV; a Randomised Crossover Trial in Patients With Acute Exacerbation of Chronic Respiratory Failure
Brief Title: Autotitrating Versus Standard Non-invasive Ventilation (NIV) in Acute Exacerbation of Respiratory Failure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty recruiting
Sponsor: ResMed (Industry)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 10/H0808/56; R&D No. 2010LF008B (Other: Research & Development Department, RBH); CI/2010/0027 (Other: Medicines & Healthcare Products Regularoty Agency (devices))
Record Dates: First submitted 2010-08-02; First posted 2010-08-03 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Respiratory Failure; Neuromuscular Disease; Chest Wall Disorder; Chronic Obstructive Pulmonary Disease; Obesity Hypoventilation Syndrome
Keywords: Acute exacerbation; Respiratory insufficiency; Respiratory failure; Hypercapnia; Hypoventilation; Sleep; Hypoxia; Titration; Non Invasive Ventilation
MeSH Terms: conditions — Respiratory Insufficiency; Neuromuscular Diseases; Pulmonary Disease, Chronic Obstructive; Obesity Hypoventilation Syndrome; Hypercapnia; Hypoventilation; Hypoxia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- autotitrating NIV (Experimental): approximately 24 hours using autotitrating non-invasive ventilation for as many hours as possible whilst an inpatient in hospital
  Interventions: Device: AutoVPAP™
- Standard non-invasive ventilation (Active Comparator): approximately 24 hours using standard non-invasive ventilation for as many hours as possible whilst an inpatient in hospital.
  Interventions: Device: VPAPIIIST-A™

INTERVENTIONS:
Device: AutoVPAP™ — Automatically titrated non-invasive ventilator, with target gross alveolar ventilation, end expiratory positive pressure, and back up respiratory rate determined by the clinician based on height and weight. The NIV must be used for as many hours as possible over the 24 hour period but breaks for meals, physiotherapy and bathroom are allowed.
  Other Names: autotitrating variable positive airway pressure; autotitrating NIV; automatically titrating NIV
  Arms: autotitrating NIV
Device: VPAPIIIST-A™ — Standard non-invasive ventilator, with inspiratory and expiratory positive pressure determined by the healthcare professional. The NIV must be used for as many hours as possible over the 24 hour period but breaks for meals, physiotherapy and bathroom are allowed.
  Other Names: standard NIV; standard non-invasive ventilator; variable positive airway pressure; VPAP
  Arms: Standard non-invasive ventilation

SUMMARY:
The aim of the study is to compare the efficacy and tolerance of autotitrating non-invasive ventilation (NIV) versus standard NIV in patients admitted to hospital with acute exacerbation of chronic respiratory failure.

The investigators hypothesise that autotitrating NIV will ventilate patients with acute exacerbations of chronic respiratory failure as effectively as standard NIV.

DETAILED DESCRIPTION:
The aim of the study is to compare the effect of two types of noninvasive ventilator (a small machine that assists breathing) in patients admitted to hospital with a sudden worsening of their existing breathing insufficiency, including an increase of carbon dioxide in the blood (hypercapnia) and acidity of the blood. Noninvasive ventilation (NIV) is standard therapy for patients with acute hypercapnic exacerbations (sudden worsening of existing breathing insufficiency) of both chronic obstructive pulmonary disease (COPD) and nonCOPD patients.

The most common type of NIV is bilevel pressure support which assists patient breathing by delivering different levels of air pressure during inspiration and expiration via a mask covering the nose or nose and mouth. Standard bilevel NIV (VPAP™) has been further developed to create a new automatically adjusting NIV (AutoVPAP™). Automatically adjusting NIV varies the inspiratory air pressure according to the airflow rates generated by the patient. This may improve patient comfort, hours of NIV use and recovery time.

Patients over the age of 18 admitted to Royal Brompton Hospital respiratory ward will be considered for entry into this randomised crossover study. If eligible for inclusion and willing to take part patients will be setup on automatically adjusting NIV or standard NIV, assigned in random order. After 24 hours on the first NIV the patient will be swapped to the alternative NIV for a further 24 hours of treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted or transferred to Royal Brompton Hospital with acute exacerbation of chronic respiratory failure, or inpatients who suffer a deterioration in respiratory status, defined as 7.25 < pH < 7.35, PaCO2 > 6.0kPa, and respiratory rate > 20bpm

Exclusion Criteria:

* < 18 years old
* pH < 7.25
* need for immediate intubation
* uncontrolled cardiac failure
* hypotensive (systolic blood pressure < 90mmHg)
* acute myocardial infarction
* acute dysrhythmia
* other system failure (e.g. acute renal failure, liver failure)
* moderate or severe bulbar weakness
* inability to understand rationale and/or consent form for study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2011-03-01 (Actual); Study Completion 2011-05-10 (Actual)

PRIMARY OUTCOMES:
pH at 1+ hour | 1 hour
  pH of arterial blood after 1 hour of treatment with non-invasive ventialtion compared baseline value

SECONDARY OUTCOMES:
pH at 4+ hours | 4+ hours of NIV treatment
  pH of arterial blood after 4 hours of treatment with non-invasive ventialtion compared to baseline value
Respiratory Rate at 1+ hour | 1+ hour of NIV treatment
  Respiratory rate after 1 hour of treatment with non-invasive ventilation compared to baseline value
Respiratory rate at 4+ hours | 4+ hours of NIV treatment
  Respiratory rate after 4 hours of treatment with non-invasive ventilation compared to baseline value
overnight mean transcutaneous carbon dioxide | 24 hours
  mean overnight transcutaneous carbon dioxide during sleep period
PaCO2 at 1+ hours | 1+ hours of NIV treatment
  Carbon dixoide level of arterial blood after 1 hour of treatment with non-invasive ventilation compared to baseline
PaCO2 at 4+ hours | 4+ hours of NIV treatment
  Carbon dioxide level in arterial blood after 4 hours of treatment with non-invasive ventilation compared to baseline value
PaO2 at 1+ hour | 1+ hour of NIV treatment
  Oxygen level in arterial blood after 1 hour of treatment with non-invasive ventilation compared to baseline value
PaO2 at 4+ hours | 4+ hours of NIV treatment
  Oxygen level in arterial blood after 4+ hours of treatment with non-invasive ventilation compared to baseline value

CONTACTS AND LOCATIONS:
Overall Officials: Anita Simonds, MD, FRCP, Principal Investigator — Royal Brompton & Harefield Hospital NHS Trust
Locations (1):
- Royal Brompton Hospital, London, United Kingdom